CLINICAL TRIAL: NCT06513702
Title: The Effectiveness of Transesophageal Lung Ultrasound (TELUS) Guided Recruitment Maneuver to Reduce Lung Atelectasis After Cardiac Surgery: a Randomized Controlled Trial
Brief Title: To Determine the Effectiveness of Transesophageal Lung Ultrasound Guided Recruitment Maneuver in Cardiac Surgery
Acronym: TELUS-REM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSCH ID-24-03856-CTF
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Bypass Surgery

STUDY DESIGN:
Intervention Model Description: This is a single center,prospective, a randomized controlled trial (RCT) study in cardiac surgery patient.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recruitment maneuver group (Experimental): Participant received TELUS guided lung reinflation during CPB weaning and TELUS guided recruitment maneuver during sternal wiring
  Interventions: Procedure: Transesophageal lung ultrasound (TELUS) guided recruitment maneuver
- Control group (Active Comparator): Participant received manual bag lung inflation during CPB weaning
  Interventions: Other: Manual bag lung reinflation

INTERVENTIONS:
Procedure: Transesophageal lung ultrasound (TELUS) guided recruitment maneuver — 1. Lung reinflation guided by transesophageal lung ultrasound (TELUS) after cardiopulmonary bypass weaning
  2. TELUS guided recruitment maneuver with continuous positive pressure of 30cmh20 for 20 seconds and 40cmh20 for 20 seconds during sternal wiring
  Arms: Recruitment maneuver group
Other: Manual bag lung reinflation — After weaning of CPB, Lung will be reinflated by 5 deep manual bag infaltion until full inflation observed by the anesthetist.
  During sternal wiring, Lung ultrasound will be examine - LUNG ultrasound score will be taken- no recruitment maneuver will be done in this contro group (Basically this group of patient is a routine practice in cardiac surgery
  Arms: Control group

SUMMARY:
This study is to evaluate the effectiveness of Transesophageal Lung ULtrasound (TELUS) guided recruitment maneuver to reduce lung atelelectasis in cardiac surgery. This is a RCT trial involving a cardiac patient that requiring used of cardiopulmonary bypass machine intraoperatively. These patient will be randomized into either intervention group or control group.

DETAILED DESCRIPTION:
Post operative pulmonary complications is a common cause of morbidity and mortality in cardiac surgery. Lung atelectasis (collapse) contributes to dysfunctional of right ventricular performance post cardiac surgery, due to increase impedance in right ventricular outflow tract. Recruitment (Lung re-expansion) maneuver is proven to be effective to reverse this effect, however it is not routinely done intraoperatively. In this study , we are conducting a randomized controlled trial to evaluate effectiveness of transesophageal lung ultrasound (TELUS) guided recruitment maneuver to reduce incidence of lung atelectasis in cardiac surgery. By this intervention, we hope that it will lead to reduce the incidence of postoperative pulmonary complications after undergoing cardiopulmonary bypass surgery.

This is a single center,prospective, a randomized controlled trial (RCT) study in cardiac surgery patient.

Patient will be randomized into 2 groups after consented into this study. After the operating list has been confirmed, we will visit the patients to be recruited, explain the purposes of this study, and then offer them to participate in this study. If the patients agree to participate in this study, they will need to sign a consent form in Malay or English language. Each participant will be assigned a code number to protect their confidentiality and the code number will be written clearly on an opaque envelope. The opaque envelope will contain participant's consent form, patient information sheet, and data collection sheet. Patient will be randomized by computer generated system into control group (group C) and recruitment maneuver group (group RM).

On the day of operation, the operation will be proceeded under general anesthesia as per standard practice. Induction and maintenance of anesthesia will be conducted as per standard practice.

Standard arterial and central venous catheterization will be inserted in all patients. The operation will be proceeded as per usual practice. The patient will be put on cardiopulmonary bypass (CBP) machine as per usual practice and the operation will be done as per scheduled. Mechanical ventilator will be suspended during CBP. Once CBP was disconnected, lung will be reinflated by giving five deep manual bag insufflations until full lung expansion observed by anaesthetist, however in interventional group lung inflation is guided by transesophageal lung ultrasound. During sternal wiring approximately about 30 minutes before the end of surgery, in interventional group they will receive a lung recruitment maneuver by continuous CPAP at 30cmH2o for 20seconds followed by PEEP 0f 8cmH20. In both groups, lung ultrasound and heart ultrasound (TOE) will be done to evaluate lung and heart function. Further assessment will be done in RM group with lung and heart ultrasound to look for changes after lung recruitment maneuver. If there is still evidence of lung collapse in the second assessment, repeated lung recruitment maneuver will be done with continuous CPAP at 40cmh20 for 20 seconds. The lung recruitment maneuver will be immediately stopped if there were signs of hypovolaemia, impairment in right ventricular contraction or a change at least 15% of baseline MAP and HR or desaturation.

Once operation is completed, patients will be reassessed again by heart ultrasound. The patient then will be transferred to the Cardiac Intensive Care Unit (CICU). The patient will be wean off from mechanical ventilator once condition permitted.

After surgery, the investigator will assess patients daily to obtain the clinical data. The patient then will be continued to be follow up until the day of discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 70 years old.
2. Elective cardiac surgery that requires used of transoesophageal ECHO.
3. New York Heart Association class I or II or III
4. Preoperative LV ejection fraction >40%
5. European System for Cardiac Operative Risk Evaluation (Euroscore) 1-6

Exclusion Criteria:

1. Pregnancy
2. Contraindication to transoesophageal ECHO - oesophageal tumour, stricture, diverticulum, or recent oesophageal or gastric surgery
3. Previous lung surgery/ history of lung radiation for cancer
4. Severe obstructive/ restrictive lung disease- Examples: Patient with home CPAP, frequent hospitalization and ICU admissions due to lung disease
5. BMI <20, > 35
6. Patient needed for re-do surgery.
7. Patient on ventricular assist device.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of lung atelectasis intraoperatively after TELUS guided recruitment | intraoperatively
  assessed by TOE during sternal wiring after recruitment maneuver

SECONDARY OUTCOMES:
Severity of Postoperative pulmonary complications. | 30 days
  Grade 0 - Absence of any complications Grade 1 - Cough, dry
  * Microatelectasis: abnormal lung findings and temperature > 37.5°C without other documented cause; normal CXR Grade 2 - Cough, productive
  * Bronchospasm
  * Hypoxemia (SpO2 ≤ 90%) at room air
  * Atelectasis: gross radiological confirmation plus either temperature > 37.5°C or abnormal lung findings
  * Hypercarbia (PaCO2 > 50 mmHg), requiring treatment Grade 3 - Pleural effusion, resulting in thoracentesis
  * Pneumonia- requiring change of antibiotic
  * Pneumothorax
  * Noninvasive ventilation- Re-intubation , with period of ventilator dependence (non-invasive or invasive ventilation) ≤ 48 hours Garde 4 - Ventilatory failure: postoperative ventilator dependence exceeding 48 hours, or reintubation with ventilator dependence exceeding 48 hours Grade 5 Death before hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mohd Fitry bin Zainal Abidin, Principal Investigator — Consultant Anaesthesiologist Universiti Malaya Medical Center

IPD SHARING:
Plan to Share IPD: Yes
By request
Supporting Information: Study Protocol
Time Frame: after 1 year
Access Criteria: through email